CLINICAL TRIAL: NCT04253912
Title: A Phase 2, Double-Blind, Randomized, Parallel Group, Placebo-Controlled, Study to Evaluate Topical 2% Povidone-Iodine Gel (VBP-245) in Subjects With Verruca Vulgaris
Brief Title: Topical 2% Povidone-Iodine Gel in Verruca Vulgaris
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Veloce BioPharma LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: VBP-245-WART2A
Record Dates: First submitted 2020-01-31; First posted 2020-02-05 (Actual); Last update posted 2021-04-01 (Actual); Status verified 2021-03

CONDITIONS: Warts
MeSH Terms: conditions — Warts

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- VBP-245 (Experimental): Topical 2% Povidone-Iodine Gel
  Interventions: Drug: VBP-245
- Control (Placebo Comparator): Placebo Gel (no Povidone-Iodine)
  Interventions: Drug: Placebo Gel (no Povidone-Iodine)

INTERVENTIONS:
Drug: VBP-245 — 2% Povidone-Iodine Gel
  Arms: VBP-245
Drug: Placebo Gel (no Povidone-Iodine) — Placebo Gel (no Povidone-Iodine)
  Arms: Control

SUMMARY:
This is a multi-center, randomized, double-blind, placebo-controlled phase 2 study in subjects 8 years of age and older who present with verruca vulgaris (common warts) and desire treatment. Subjects may have up to a total of 6 common warts located on their trunk or extremities that will be treated with study medication and followed throughout the study protocol therapy. All warts will be treated two times per day (BID) for12 weeks. Approximately 90 subjects will be enrolled in this study.

ELIGIBILITY:
Inclusion Criteria:

* Subject is able to comprehend and is willing to sign an informed consent/assent for participation in this study.
* Male or female ≥ 8 years old.
* Subject has a clinical diagnosis of verruca vulgaris (common warts).
* Subject has up to 6 warts located on the trunk or extremities

Exclusion Criteria:

* Subject has clinically atypical warts on the trunk or extremities.
* Subject is immunocompromised (e.g., due to chemotherapy, systemic steroids, genetic immunodeficiency, transplant status, etc.)
* Subject has periungual, subungual, genital, anal, mosaic, plantar, flat, or filiform wart identified as a wart for study treatment.

Min Age: 8 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2020-02-12 (Actual); Primary Completion 2021-01-05 (Actual); Study Completion 2021-04 (Estimated)

PRIMARY OUTCOMES:
Decrease in wart diameter (mm) | 12 weeks

SECONDARY OUTCOMES:
Resolution of wart | 12 weeks
  Wart diameter = 0 mm
Application Site Reaction Adverse Events | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Barone, MD, Study Director — Veloce BioPharma LLC
Locations (7):
- United States (7):
  - Veloce BioPharma Clinical Trial Site, Hunt Valley, Maryland
  - Veloce BioPharma Clinical Trial Site, Plymouth Meeting, Pennsylvania
  - Veloce BioPharma Clinical Trial Site, Sugarloaf, Pennsylvania
  - Veloce BioPharma Clinical Trial Site, Upper Saint Clair, Pennsylvania
  - Veloce BioPharma Clinical Trial Site, Fort Mill, South Carolina
  - Veloce BioPharma Clinical Trial Site, Arlington, Virginia
  - Veloce BioPharma Clinical Trial Site, Lynchburg, Virginia

IPD SHARING:
Plan to Share IPD: Undecided
Aggregate data will be shared with study investigators.